CLINICAL TRIAL: NCT04957875
Title: Timing of Endoscopy for Acute Variceal Bleeding in Patients With Cirrhosis (CHESS1905): a Nationwide Cohort Study
Brief Title: Timing of Endoscopy for Acute Variceal Bleeding in Patients With Cirrhosis
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing 302 Hospital (Other); Tianjin Third Central Hospital (Other); The Sixth People's Hospital of Shenyang (Other); Shanxi Bethune Hospital (Other); Linyi People's Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Institute of Portal Hypertension, The First Hospital of Lanzhou University, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS1905
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cirrhosis, Liver; Portal Hypertension; Varice Bleed
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- urgent endoscopy group: endoscopy <6h after admission
  Interventions: Device: emergency endoscopic therapy
- early endoscopy group: endoscopy 6-24h after admission
  Interventions: Device: emergency endoscopic therapy

INTERVENTIONS:
Device: emergency endoscopic therapy — When cirrhotic patients presented with AVB to the emergency department, emergency physicians consulted gastroenterologists on duty to assess the patient for suitability for endoscopy, usually after initial stabilization. Performance of endoscopy and its timing was at the discretion of the gastroenterologist on call. Therapeutic endoscopy for AVB was performed within 24 hours after consultation by an experienced attending endoscopist, using standard forward-viewing upper gastrointestinal video endoscopes at individual centers. Written informed consent for endoscopy was obtained before each procedure. The standard of care at all hospitals was to administer a vasoactive agent and antibiotics upon the patient's presentation. Packed red blood cells were transfused at the discretion of the attending gastroenterologist.

SUMMARY:
Cirrhotic patients with AVB across 34 university medical centers in 30 cities in China from February 2013 to May 2020 who underwent endoscopy within 24 hours were included in this study. Patients were divided into an urgent endoscopy group (endoscopy <6h after admission) and an early endoscopy group (endoscopy 6-24h after admission). Outcomes included the incidence of 5-day rebleeding, in-hospital mortality, need for intensive care unit (ICU) and the length of hospital stay after the endoscopy management. Multivariable analysis was performed to identify risk factors for rebleeding. A propensity score matching (PSM) analysis was performed to achieve a balance at baseline between the urgent and early groups.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of cirrhosis (based on liver biopsy or the combination of clinical, biochemical, and imaging findings)
* witnessed or reported evidence of gastrointestinal haemorrhage (hematemesis, melenemesis, or hematochezia)
* esophageal or gastric varices confirmed endoscopically as the source of bleeding

Exclusion Criteria:

* severe dysfunction of a major extrahepatic organ (e.g., heart failure, pulmonary disease, and terminal malignancy except hepatocellular carcinoma)
* history of endoscopic therapy for varices (ligation or sclerotherapy) within three months
* incomplete or missing data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complete demographic and clinical data of patients with cirrhosis associated with AVB who underwent emergency endoscopy within 24 hours between February 2013 and May 2020 across 34 university hospitals from 30 cities in China was retrospectively reviewed. Two independent investigators (Liu C and Huang Y) reviewed the medical records, including demographic, laboratory, clinical and endoscopic data.
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
the incidence of 5-day rebleeding after emergency endoscopy | 6 months

SECONDARY OUTCOMES:
the in-hospital mortality | 6 months
need for ICU | 6 months
the length of hospital stay | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Lanzhou university, Lanzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Background] Lau JYW, Yu Y, Tang RSY, Chan HCH, Yip HC, Chan SM, Luk SWY, Wong SH, Lau LHS, Lui RN, Chan TT, Mak JWY, Chan FKL, Sung JJY. Timing of Endoscopy for Acute Upper Gastrointestinal Bleeding. N Engl J Med. 2020 Apr 2;382(14):1299-1308. doi: 10.1056/NEJMoa1912484. PMID 32242355
- [Background] Chen PH, Chen WC, Hou MC, Liu TT, Chang CJ, Liao WC, Su CW, Wang HM, Lin HC, Lee FY, Lee SD. Delayed endoscopy increases re-bleeding and mortality in patients with hematemesis and active esophageal variceal bleeding: a cohort study. J Hepatol. 2012 Dec;57(6):1207-13. doi: 10.1016/j.jhep.2012.07.038. Epub 2012 Aug 8. PMID 22885718